CLINICAL TRIAL: NCT02185196
Title: Vitamin D Supplementation: Impact on Severe Pneumonia Among Under-five Children
Brief Title: Vitamin-D Supplementation: Impact on Severe Pneumonia Among Under-five Children
Acronym: Vitamin-D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-13088
Record Dates: First submitted 2014-06-22; First posted 2014-07-09 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-02

CONDITIONS: Pneumonia
Keywords: Vitamin D,; Severe pneumonia,; Under-five children,; Randomised; Controlled; Trial (RCT); Morbidity
MeSH Terms: conditions — Pneumonia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Active Comparator): Vitamin D3, Doses form: 20,000 IU vitamin D3 in children <6 months, 50,000 IU in children 6-12 months and 1,00,000 IU in children 13-59 months of age on first day and thereafter 10,000 IU for next 4 days.
  Interventions: Drug: Vitamin D3
- Miglyol-oil (Placebo Comparator): 20,000 IU Miglyol-oil in children <6 months, 50,000 IU in children 6-12 months and 1,00,000 IU in children 13-59 months of age on first day and thereafter 10,000 IU for next 4 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — 20,000 IU vitamin D3 in children <6 months, 50,000 IU in children 6-12 months and 1,00,000 IU in children 13-59 months of age on first day and thereafter 10,000 IU for next 4 days
  Other Names: Vigantol-oil
  Arms: Vitamin D3
Drug: Placebo — 20,000 IU Miglyol-oil in children <6 months, 50,000 IU in children 6-12 months and 1,00,000 IU in children 13-59 months of age on first day and thereafter 10,000 IU for next 4 days
  Other Names: Miglyol Oil
  Arms: Miglyol-oil

SUMMARY:
Background:

* Burden: Pneumonia is the leading cause of morbidity and mortality in under-five children, particularly in developing countries.
* Knowledge gap: Although many studies have reported an association between vitamin D deficiency and pneumonia, there is lack in information on its therapeutic impact, i.e. the impact of vitamin D supplementation in the management of childhood pneumonia.
* Relevance: Vitamin D plays an important role in modulating the innate immune response against infections. We, therefore, propose to conduct this study to assess the impact of vitamin D supplementation, in addition to standard antibiotic and supportive therapy, on the outcome of severe childhood pneumonia.

Hypothesis: The investigators hypothesise that in the management of hospitalized severe pneumonia in under-five children, vitamin D3 supplementation, as an adjunct to the standard antibiotic and other supportive therapy, will hasten recover from severe pneumonia and may thereby shorten duration of severe pneumonia and also reduce the risk of new episode of pneumonia.

Objectives: The objective of the investigators study is to assess the clinical benefit of oral supplementation of vitamin D3, in addition to standard antibiotic and other supportive therapy, to hospitalised, under-five children with severe pneumonia.

Methods: This would be a randomised, double blind, controlled clinical trial (RCT). Children of either sex, aged 3-59 months, attending the Dhaka Hospital of icddr,b, with clinically diagnosed severe pneumonia will comprise the study population. Eligible children will be allotted a sequential study number, which will have been previously assigned to vitamin D or placebo in accordance with the randomisation. The study staff and mothers/ caregivers of the children will be blinded as to whether vitamin D3 or placebo has been added to their child's diet. Infants aged 3-5 months will receive breast milk and/or infant formula, and those 6 months or older will receive "Milk Suji" as a complementary food. Vitamin D3 supplementation will be given on five consecutive days, from the day of enrolment in addition to standard antibiotic and other supportive therapy.

Outcome measures/variables:

Primary outcome measure will be time to resolution of severe pneumonia.

Secondary outcome measures will be duration of hospitalization, fever, tachypnoea, chest in drawing, hypoxia, lethargy and inability to feed during hospital stay and as well as new episode of pneumonia after discharge.

DETAILED DESCRIPTION:
Hypothesis to be tested:

In a hypothesis testing research proposal, briefly mention the hypothesis to be tested and provide the scientific basis of the hypothesis, critically examining the observations leading to the formulation of the hypothesis.

Does this research proposal involve testing of hypothesis: 0 No 1 Yes (describe below)

The investigators hypothesise that supplementation of vitamin D3 (Cholecalciferol), in addition to standard antibiotic and other supportive therapy in the management of under-five children with severe pneumonia will significantly shorten the duration of severity of pneumonia and thereby reduce hospital stay and also reduce the risk of new episode of pneumonia.

Specific Objectives:

Objective: To assess the clinical benefit of oral vitamin D3 supplementation, in addition to standard antibiotic and other supportive therapy, in the management of hospitalised, under-five children with severe pneumonia.

Primary objective: To compare the duration of severe pneumonia of children in the two study groups receiving the standard therapy (appropriate antibiotic and other supportive therapy) with those receiving vitamin D supplementation in addition to the standard therapy.

Secondary objectives:

* To compare the duration of hospitalization, fever, tachypnoea, chest in drawing, hypoxia, lethargy and inability to feed during hospital stay, in under-five children in the two study groups, as mentioned under the primary aim.
* To compare the recurrence of new episode of pneumonia over the next 6 months after discharge from hospital in the two study groups.
* To identify the optimum safety dose of vitamin D3 for different groups of under-five children.
* In severe pneumonia patient who also have acute watery diarrhoea we will assess the indirect absorption of vitamin D by measuring serum vitamin D level and will also assess the clinical outcome in the subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged 3 - 59 months, with a clinical diagnosis of severe pneumonia with or without diarrhea.

Exclusion Criteria:

1. Known case of hypercalcaemia or allergy to vitamin D, as determined by history or previous medical records.
2. Congenital Heart disease, evidenced by clinical exam or past medical records.
3. Renal or hepatic insufficiency, evidenced by clinical exams or past medical records.
4. Known case of tuberculosis, evidenced by medical records
5. Known case of asthma, evidenced by history and clinical exam findings.
6. Critically ill children requiring ICU care, such as those with septic shock or cardiac arrest or apnoea.
7. Received vitamin D or calcium supplementation within the last 4 weeks before current admission, as evidenced by history or medical prescription.
8. Any children diagnosed as hypernatraemia during the main phase of the study.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Time taken for recovery from severe pneumonia | 12 months

SECONDARY OUTCOMES:
Duration of hospitalization | 12 months
Time taken for normalisation of temperature | 12 months
Time taken for normalisation of respiratory rate | 12 months
Time taken for recovery from chest in drawing | 12 months
Time taken for oxygen saturation to normalise | 12 months
Time taken for normalization of mental status | 12 months
Time taken for normalization of child feeding | 12 months
Proportion of study children who will develop new episode of pneumonia during the follow up period | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fahmida Chowdhury, MBBS, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital of the International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Chowdhury F, Shahid ASMSB, Tabassum M, Parvin I, Ghosh PK, Hossain MI, Alam NH, Faruque ASG, Huq S, Shahrin L, Homaira N, Hassan Z, Akhtar Z, Mah-E-Muneer S, Fuchs GJ, Ahmed T, Chisti MJ. Vitamin D supplementation among Bangladeshi children under-five years of age hospitalised for severe pneumonia: A randomised placebo controlled trial. PLoS One. 2021 Feb 19;16(2):e0246460. doi: 10.1371/journal.pone.0246460. eCollection 2021. PMID 33606713